CLINICAL TRIAL: NCT03749967
Title: Developing a Novel rTMS Intervention for Transdiagnostic Psychosocial Rehabilitation: A Dose Finding Study
Brief Title: rTMS for Emotional Difficulties in Verterans
Acronym: rTMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2886-P; RX002886 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Mental Health; Depression; rTMS; Anxiety; PTSD; Psychosocial Impairment
Keywords: Depression
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Veterans will be randomized to 10 different doses of accelerated intermittent theta burst rTMS for remediation of transdiagnostic psychosocial impairment. The goal is to determine the optimal dose in terms of efficacy while minimizing burden and side effects.
Who Masked: Participant
Masking Description: All participants will be randomized to 10 different active doses of accelerated, intermittent theta burst rTMS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (10):
- Dose 1 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is five sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 2 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 2 is ten sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 3 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is fifteen sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 4 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is twenty sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 5 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is twenty-five sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 6 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is thirty sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 7 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is thirty-five sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 8 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is forty sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 9 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is forty-five sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 10 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is fifty sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — MagVenture MagPro TMS System would be utilized to deliver 3-minute sessions of intermittent theta burst to left dorsolateral prefrontal cortex.

SUMMARY:
Mental illness rarely occurs as a single, easily categorized condition. Instead, multiple disorders often co-occur. This complicates the treatment plan for many Veterans, especially those suffering the most severe dysfunction. This also means that clinical research aimed at one specific disorder may not be optimized to treat the realworld presentation of neuropsychiatric illness. The investigators propose in this study to develop a novel, non-invasive brain stimulation treatment that would promote rehabilitation for Veterans suffering a wide range of emotional difficulties. More specifically, the investigators propose to up-regulate the brain circuitry that supports flexible problem solving and contending with daily demands. Rather than focusing on reducing the symptoms of a specific disorder to reduce the intrusion into daily life, the investigators propose to augment those brain circuits that promote adaptive cognition and thus quality of life.

DETAILED DESCRIPTION:
The investigators propose that because rTMS to dlPFC is targeting cognitive neurocircuitry integral to adaptive cognitive functioning, promoting neuroplasticity in this network with rTMS could be more precisely optimized to improve quality of life across psychosocial domains and across neuropsychiatric presentations. The investigators postulate that through up-regulating cognitive control circuitry with rTMS that an individual would have 1) enhanced capacity for successfully contending with the shifting contingencies of daily life and 2) improved ability to regulate intrusive affect and impulses. As a function of these processes an individual is expected to experience reduced psychosocial impairment. Thus, the investigators propose that rather than targeting specific symptom reductions in specific disorders, rTMS could be dosed for efficacy in enhancing psychosocial functioning. Such an approach has the potential to enhance rehabilitation for far more Veterans suffering a range of neuropsychiatric conditions.

Aim 1. Establish the dose-response curve for improved psychosocial functioning secondary to accelerated rTMS in a transdiagnostic anxious and depressed sample of Veterans.

Aim 2. Establish the safety, feasibility, and acceptability of an accelerated delivery schedule of therapeutic rTMS for improved psychosocial functioning in a transdiagnostic anxious and depressed sample of Veterans.

Exploratory Aim 3. Establish whether neurocognitive function demonstrates a dose-response function to accelerated rTMS similar to psychosocial functioning in a transdiagnostic anxious and depressed sample.

Note: COVID-19 pandemic put a pause on enrollment.

ELIGIBILITY:
Inclusion Criteria:

* A negative urine pregnancy test, if female subject of childbearing potential.
* Able to speak English and complete study forms, adhere to treatment regimens, and be willing to return for regular visits.
* After full explanation of the study, willingness of participant is demonstrated by signing the informed consent form.

Exclusion Criteria:

* Clinically unstable medical disease:

  * cardiovascular
  * renal
  * gastrointestinal
  * pulmonary
  * metabolic
  * endocrine
  * other
  * CNS disease deemed progressive
  * Moderate or severe traumatic brain injury (TBI) - (using VA/DoD Clinical Practice Guidelines)
* Pregnant females or those currently breast-feeding.
* Current or history of schizophrenia or other psychotic disorder, except psychosis not otherwise specified (NOS) when the presence of sensory hallucinations is clearly related to the subject's trauma, Bipolar Type I disorder, or dementia

  * vascular
  * Alzheimer's disease
  * other types)
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) within 6 days of study entry, with the exception of alcohol use disorder, which, at the discretion of the study team, may be permitted.

  * See further explanation under protection from risk.
* Active participation or plan for enrollment in another evidence-based psychotherapeutic clinical trial

  * Participation in other psychotherapeutic modalities must have been stable for 3 months prior to enrollment and must remain stable throughout participation.
* Currently taking medications that have short half-lives, lower the seizure threshold, and do not have evidence of antidepressant efficacy. These include:

  * high dose theophylline or stimulants such as methylphenidate
  * patients taking bupropion must be on a stable dose and take less than or equal to 300 mg/day. Stable means the same dose for 5 half-lives.
* An implanted device in subject's head (shunt, cochlear implant) and/or metal in subject's head (other than dental implant).

History of seizures or a seizure disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (IPF) | 4 weeks post-treatment
  The IPF is an 80-item self-report measure used to assess functional impairment across multiple psychosocial domains of functioning. It was iteratively developed in 697 male and female Veteran stakeholders to identify relevant domains of functional impairment common in PTSD and related psychiatric dysfunction. Total score range=0-480. Increased scores pre- to 4 weeks post-treatment would indicate improved function.
World Health Organization Quality of Life - Brief Form (WHOQOL-BF) | 4 weeks post-treatment
  The WHOQOL-BREF is a 26-item self-assessment form. Questions are rated on a 5 point scale (from 1-5) Likert scale. Reflects four domains: physical, psychological, social and environment.
Illness Intrusiveness Rating Scale (IIRS) | 4 weeks post-treatment
  The IIRS is a self-report measure of the extent of psychosocial impairment secondary to illness. Total score range=13-91. Decreased scores pre- to 4 weeks post-treatment would indicate improved function.

SECONDARY OUTCOMES:
Neurocognitive performance | 4 weeks post-treatment
  Participants would complete a computerized battery, which includes well-validated computer-adaptations of neuropsychological tests. Tasks assess the following domains: information-processing speed, executive function, sustained attention/vigilance, verbal memory, working-memory capacity, inhibition/impulsivity, and sensorimotor function. Improved performance pre- to 4 weeks post-treatment would indicate improved function.
Inventory of Depression and Anxious Symptoms (IDAS-II) | 4 weeks post-treatment
  Questions are rated on a scale from 1-5 and covers a wide array of psychological measures
Hamilton Scale for Depression (HAM-D) | 4 weeks post-treatment
  Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. 10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Mood and Anxiety Symptom Questionnaire (MASQ) | 4 weeks post-treatment
  Questions designed to assess symptoms of general distress using a 5-point Likert scale ranging from 1"not at all" to 5 "extremely".

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. McTeague, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No